CLINICAL TRIAL: NCT06138366
Title: The Effect of Foot-Ankle Characteristics, Lower Extremity Muscle Strength, Walking Speed and Functional Exercise Capacity on Kinesiophobia in Elderly Individuals: A Three-Center Observational Study
Brief Title: Factors Affecting Kinesiophobia in the Elderly
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Ayşe Toraman, Lecturer, Bulent Ecevit University
Other Study IDs: AYSE TORAMAN KARAGULMEZ2
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Aged
Keywords: Kinesophobia; Aged; Walking speed; foot
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In epidemiological studies, the incidence of foot problems has been found to be high as a result of the increase in life expectancy. The changes that occur in the foot with advancing age are extremely important in that they affect how the foot functions and transfer these effects to other body systems while standing and walking. These changes can also cause foot pain, limit mobility, impair functional performance in activities where the foot bears weight, and increase the risk of falling. In recent years, the level of kinesiophobia in elderly individuals; It seems to attract attention in terms of its effects on balance, falling, risk of falling, fear of falling, depression, physical activity level and quality of life. However, in the elderly living in nursing homes; It is not yet known how ankle joint position sense, foot posture, pain, foot-ankle disability, activity limitation, lower extremity muscle strength, walking speed and functional exercise capacity affect kinesiophobia. By elucidating these relationships, it will be possible to develop intervention strategies aimed at increasing foot-ankle characteristics, lower extremity muscle strength, walking speed and functional capacity, which are modifiable risk factors. The aim of this study is to examine the relationship between kinesiophobia and foot-ankle characteristics, lower extremity muscle strength, walking speed and functional exercise capacity in elderly people living in nursing homes.

DETAILED DESCRIPTION:
The research will be carried out in Zonguldak Center, Karadeniz Ereğli İzmirlioğlu and Çaycuma Nursing Homes affiliated with the Zonguldak Provincial Directorate of Family and Social Services. Among the elderly individuals staying here, those who are volunteers and meet the inclusion criteria will be included in the study.The study will begin after receiving ethics committee approval. After the ethics committee permission of the study is obtained by the researchers, the necessary permissions to conduct this study will be obtained by applying to the Zonguldak Provincial Directorate of Family and Social Services. Data collection by researchers will begin after receiving permission from the relevant units.Before starting the evaluations on elderly individuals within the scope of the study, all elderly individuals will be given all necessary information about the purpose and procedure of the study by the researchers and they will sign an informed consent form.Permission will be requested by the researchers from all test and scale owners for all tests and scales that the researchers will use in the study.

The study was planned as a cross-sectional observational study. In the study, the sample size was calculated with G-Power and a power analysis was performed.The sample size required for the study is 64, and the minimum number of people that will provide 80% test power and 95% confidence level is 64, with effect size = 0.3 for Pearson correlation analysis.This sample width also includes the sample widths required for other analysis methods to be used within the scope of the study. The relevant calculation was made in the G-Power 3.1.9.2 package program.In the study, the relationships between the kinesiophobia status of elderly individuals and the variables of foot-ankle characteristics, lower extremity muscle strength, walking speed and functional exercise capacity will be examined. In addition, according to the kinesiophobia levels of elderly individuals, the cut-off value is taken as 37 points and the score is; Those with a score below 37 points will be grouped as individuals with low kinesiophobia, and those with a score of 37 points and above will be grouped as individuals with high kinesiophobia, and the relationships between the variables will be analyzed.

The research is planned to be carried out by the researchers in Zonguldak Center, Kdz.Ereğli İzmirlioğlu and Çaycuma Nursing Homes between 9 December 2023 and 31 December 2024. As Evaluation Methods; For socio-demographic status, Demographic Information Form, for evaluation of foot deformities and problems; Foot deformity and problems evaluation form, for disease status, Charslon Comorbidity Score, for cognitive status; Standardized Mini Mental State Test, for fall risk and balance assessment; Timed Up and Go Test for walking speed; 10-meter Forward Walk Test, 3-meter Backward Walk Test for functional capacity evaluation; Six Minute Walk Test, for assessment of dyspnea and fatigue severity; Modified Borg Scale, for evaluation of foot-ankle characteristics; Ankle Joint Position Sense Assessment, Foot Posture Index, Foot Function Index, for lower extremity muscle strength; Sit-Stand Chair Test for fear of movement; Tampa Kinesiophobia Scale will be used. Within the scope of the study, participants' joint position sense will be evaluated with "Universal Goniometer", walking speed with "Digital Stopwatch" and blood pressure with "Sphygmomanometer (Omron M3 HEM-7155-E)".

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years of age and older
* Stay in a nursing home
* Getting a score of 24 or higher on the Standardized Mini Mental State Test
* Being able to walk with a cane or without a cane
* Know how to read and write

Exclusion Criteria:

* Being vision problem that cannot be corrected with glasses or lenses
* Being hear problem that cannot be corrected with hearing aids
* Being blood pressure unsafe for exercise (>180/100 or <100/60 mmHg at rest)
* Being severe respiratory and cardiac problems
* History of lower extremity surgery in the last six months
* Being severe orthopedic and neurological deficits that may affect walking
* History of recurrent falls (more than one fall in the last year)
* Being do exercise more than 150 minutes a week
* Participating in any exercise program in the last six months
* Have received any foot health treatment in the last six months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Volunteer elderly individuals living in Zonguldak Center, Karadeniz Ereğli İzmirlioğlu and Çaycuma Nursing Homes affiliated with the Zonguldak Provincial Directorate of Family and Social Services and individuals who meet the inclusion criteria will participate in the research. In order to conduct the research, an application will be made to Zonguldak Provincial Directorate of Family and Social Services for the necessary permissions and permissions will be obtained. All individuals who volunteer to participate in the study will be given all necessary information about the purpose and procedure of the study before starting the study. All volunteers will then need to sign an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Foot Posture | Baseline
  Foot Posture İndex: The test score is calculated by assigning values between -2 and +2 to the 6 criteria on the foot and summing the scores from all criteria.
  A test score of 0 indicates that the foot is in a neutral position. A positive test score indicates standing pronation. A negative test score indicates standing supination.
Foot Function | Baseline
  Foot Function İndex:The scale consists of three subscales: pain, disability, and activity limitation. There are 23 questions in total. The participants are asked to score all questions with a visual analog scale scaled between 0-10, taking into account their foot condition in the last week. To calculate the sub-scales and the total score, the score of each item is added, divided by the sum of the maximum scores of the items and multiplied by 100. Higher scores indicate more pain, disability, and activity limitation.
Ankle Joint Position Sense | Baseline
  Individuals will be asked to bring their neutral feet to the desired target positions (10 degrees of dorsiflexion, 10 degrees of plantar flexion, 20 degrees of plantar flexion). Measurements will be repeated 3 times for each target angle. The absolute value of the deviations from the target angles will be recorded and the average of the deviations occurring during the 3 repetitions will be taken.
Lower extremity muscle strength | Baseline
  Sit-Up Chair Test: The number of times the individual sits and stands in a chair during 30 seconds will be recorded as the individual's score.
Forward Walking Speed | Baseline
  10 meters Forward Walk Test:The time it takes to cover the ten meters at the person's normal speed will be recorded. The test is performed twice, and the average value is recorded in meters/second with the stopwatch.
Backward Walking Speed | Baseline
  3 meters Backward Walk Test:The time taken for the person to walk backwards as fast as possible will be recorded. The test is performed once and its duration is recorded in meters/second with a stopwatch.
Kinesiophobia | Baseline
  Tampa Kinesiophobia Scale:Responses on the Tampa Kinesiophobia Scale are classified as strongly disagree, disagree, agree and strongly agree. There are two types of expressions (direct and inverse) in the scale. While these expressions are scored, those who get 1 point turn into 4, and those who get 4 points turn into 1.4-point answers in direct statements indicate a high level of kinesiophobia. In reversed expressions, answers with a value of 1 indicate a high level of kinesiophobia, and answers with a value of 4 indicate a low level of kinesiophobia. Scores from the scale range from 17 to 68. The score obtained from the scale constitutes the individual's score that should be interpreted at the level of kinesiophobia. A high score indicates a high level of kinesiophobia.
Functional Exercise Capacity | Baseline
  Six-minute walk test: The distance traveled will be measured by walking in a straight 30-meter corridor for six minutes. More distance traveled indicates better functional capacity.

SECONDARY OUTCOMES:
Balance Performance | Baseline
  In the test, the person will be asked to get up from his chair, walk 3 meters at a safe and normal speed, turn, walk back and sit on the chair.
  The time required by the individual to perform this movement will be recorded in seconds (sec). Three repetitions will be made, the average will be taken and the result will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: AYŞE TORAMAN KARAGÜLMEZ, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Zonguldak Center, Kdz. Ereğli İzmirlioğlu and Çaycuma Nursing Homes, Zonguldak, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No